CLINICAL TRIAL: NCT00039117
Title: A Phase I Study of G3139 ( NSC # 683428) in Combination With Cytarabine and Daunorubicin in Previously Untreated Patients With Acute Myeloid Leukemia (AML)>= 60 Years of Age
Brief Title: Oblimersen, Cytarabine, and Daunorubicin in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01409; OSU-0164; NCI-4630; CDR0000069353; U01CA076576 (NIH)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities | interventions — oblimersen; Cytarabine; Daunorubicin

ARMS (1):
- Arm I (Experimental): INDUCTION THERAPY: Patients receive oblimersen (G3139) IV continuously on days 1-10 and cytarabine IV continuously on days 4-10. Patients also receive daunorubicin IV daily on days 4-6.
  Patients with bone marrow cellularity of at least 20% and at least 5% leukemic blasts at day 17 or evidence of refractory disease receive a second induction comprising G3139 IV continuously on days 1-8, cytarabine IV continuously on days 4-8, and daunorubicin IV on days 4-5.
  CONSOLIDATION THERAPY: Beginning no sooner than 14 days after hematologic recovery from induction therapy, patients receive G3139 IV continuously on days 1-8 and cytarabine IV over 4 hours on days 4-8. Patients receive a second course of consolidation therapy no sooner than 14 days after hematologic recovery from the first course.
  Interventions: Biological: oblimersen sodium; Drug: cytarabine; Drug: daunorubicin hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effectiveness of combining oblimersen with cytarabine and daunorubicin in treating older patients who have previously untreated acute myeloid leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Oblimersen may help cytarabine and daunorubicin kill more cancer cells by making them more sensitive to chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of daunorubicin in combination with cytarabine and oblimersen in older patients with previously untreated acute myeloid leukemia.

II. Determine the qualitative and quantitative toxic effects of this regimen in these patients.

III. Determine the pharmacokinetics of oblimersen in this regimen in these patients.

IV. Determine the disease-free survival and overall survival of patients treated with this regimen.

V. Assess the spontaneous rate of apoptosis in leukemic blasts in patients before and after initiation of treatment with oblimersen.

VI. Determine therapeutic response (complete remission) in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of daunorubicin. Patients are stratified according to disease status (primary vs secondary).

INDUCTION THERAPY: Patients receive oblimersen (G3139) IV continuously on days 1-10 and cytarabine IV continuously on days 4-10. Patients also receive daunorubicin IV daily on days 4-6.

Patients with bone marrow cellularity of at least 20% and at least 5% leukemic blasts at day 17 or evidence of refractory disease receive a second induction comprising G3139 IV continuously on days 1-8, cytarabine IV continuously on days 4-8, and daunorubicin IV on days 4-5.

CONSOLIDATION THERAPY: Beginning no sooner than 14 days after hematologic recovery from induction therapy, patients receive G3139 IV continuously on days 1-8 and cytarabine IV over 4 hours on days 4-8. Patients receive a second course of consolidation therapy no sooner than 14 days after hematologic recovery from the first course.

Cohorts of 3-6 patients receive escalating doses of daunorubicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary or secondary acute myeloid leukemia (AML)

  * More than 20% bone marrow blasts
  * Myelodysplastic syndromes (MDS) or a chronic myeloproliferative disorder antecedent to AML allowed
  * Therapy-related AML allowed
  * No acute promyelocytic leukemia
* At least 4 weeks
* Bilirubin no greater than 2 mg/dL
* ALT and AST no greater than 2 times upper limit of normal (unless directly attributable to AML)
* Creatinine no greater than 2.5 mg/dL
* Ejection fraction at least 50% by MUGA or echocardiogram
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No allergy to any of the study medications
* No other uncontrolled concurrent illness
* No serious medical or psychiatric illness that would preclude giving informed consent
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior therapy for primary AML except emergency leukapheresis
* No prior anthracyclines
* No prior chemotherapy for primary AML except hydroxyurea for hyperleukocytosis
* At least 3 months since prior chemotherapy for MDS or chronic myeloproliferative disorders antecedent to AML
* No other concurrent chemotherapy
* No concurrent corticosteroids as anti-emetics
* No concurrent steroids except for adrenal failure or septic shock
* No concurrent hormonal therapy except hormones for non-disease-related conditions (e.g., insulin for diabetes, tamoxifen or equivalent for breast cancer prevention or adjuvant treatment, or estrogens or progestins for gynecologic indications)
* No prior radiotherapy for primary AML except cranial radiotherapy for CNS leukostasis
* No concurrent palliative radiotherapy
* No concurrent whole brain radiotherapy
* No other concurrent investigational or commercial agents or therapies
* No concurrent cyclooxygenase-2 inhibitors

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-04; Primary Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
MTD of cytarabine and daunorubicin in combination with G3139, defined as the dose level just below the dose level at which DLT is observed in 2 patients, graded according to NCI CTC version 2.0 | Up to day 10
Incidence of adverse events, graded according to NCI CTC version 2.0 | Up to 2 years
  We will define the qualitative and quantitative toxicities in regard to organ specificity, time course, predictability, and reversibility.

SECONDARY OUTCOMES:
Pharmacokinetics of G3139 | During induction therapy on day 1 at hour 0 and 24hours after G3139 administration; day 4 at hour 73 before cytarabine administration; day 11 at hour 0 and .5, 1, 2, 4, 6, and 8 hours
Level of bcl-2 in circulating and/or marrow leukemic blasts before and after initiation of treatment with G3139 | Up to 18 weeks
Spontaneous rate of apoptosis in leukemic blasts before and after initiation of treatment with G3139 | Up to 18 weeks
Incidence of therapeutic response (complete remission [CR]) | Up to 2 years
Disease-free survival | Up to 2 years
Overall survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marcucci, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States